CLINICAL TRIAL: NCT00494117
Title: Investigation of Heart Failure Status Over Time Using Respiratory Parameters
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Rachel Coxon, ResMed
Other Study IDs: X07- 0052
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Heart Failure, Congestive; Sleep Apnea Syndromes
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ApneaLink — A two channel sleep screening device for the assessment of Sleep Disordered Breathing.

SUMMARY:
The purpose of the study is to investigate respiratory indicators for clinically important changes in Heart Failure status over time.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Heart Failure (as determined by Echocardiogram or by treating physician)

Exclusion Criteria:

* Malignant disease affecting gas exchange or respiratory parameters
* Medications compromising breathing with no adverse affects on heart failure
* Clinically significant (moderate to severe) asthma requiring therapy
* Chronic parenchymal lung disease (FEV1/FVC ratio = 65% or as determined by the treating physician)
* Severe pulmonary hypertension
* Heart failure due to alcohol abuse or chemotherapy
* Narcotic abuse/intravenous drug use (including HIV+ and hepatitis C)
* Alcohol consumption > 80g/day
* Patients receiving home Oxygen
* Methicillin- resistant Staphylococcus aureus infection
* Narcolepsy
* Cataplexy
* Enrolled in any concurrent study, that may confound the results of this study.
* Inability or refusal to sign the Patient Consent Form
* Inability or refusal to adhere to protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population under investigation is moderate to severe heart failure who are outpatients of a major Sydney hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Coxon, BE/MBiomedE, Study Director — ResMed/The University of New South Wales; Klaus Schindhelm, PhD, Study Director — ResMed/The University of New South Wales; Jodie Lattimore, PhD, Study Director — Royal Prince Alfred Hospital, Sydney, Australia; Ian Wilcox, PhD, Principal Investigator — Royal Prince Alfred Hospital/The University of Sydney
Locations (1):
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia